CLINICAL TRIAL: NCT04532476
Title: Effect of a Double Dose of Photobiomodulaton Therapy on Orthodonthic Pain Caused by Elastomeric Separators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vjera Perkovic, Doctor of dental medicine, orthodontist specialist, University Hospital Rijeka
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UHRijeka- laser
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Pain Relief Caused by Placing Orthodontic Separators
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a single -blinded, placebo controlled, split-mouth study. The design was split-mouth to eliminate all components related to differences among subjects.
Who Masked: Participant, Outcomes Assessor
Masking Description: It was determined in advance that the right side of the upper jaw was treated with laser, and the left side was placebo.Placebo side was treated the same way with the difference that the laser was switched off, but with the maintained sound signal, implying laser was working, so that partici-pants were blinded to the allocation of the group, only the operator knew whether the side is laser treated or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treated side (Experimental): Group of 22 participants whose mucose around right maxillary permanent molar was treated with laser.
  Interventions: Device: Low level laser therapy
- Placebo side (Placebo Comparator): Placebo side was LEFT side.It was treated the same way as right with the difference that the laser was switched off, but with the maintained sound signal, implying laser was working, so participants were blinded to the allocation of the group, only the operator knew whether the side is laser treated or placebo.
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Low level laser therapy — Diode laser (Laser HF, Hager-Werken GmbH & Co., Duisburg, Germany) was applied to the RIGHT side. Laser was set at PDT mode (660nm) acupuncture therapy. The power of the laser was set at 90 mW in intervals of 80 seconds as recommended by the manufacturer.
  The laser was applied perpendicular in contact with the mucosa on 1 point of the buccal and 1 point on the palatal side of the first molar approximately on the middle part of the root, with the 10mm distance from the laser to the mucosa. Each point was treated in 3 intervals, 80s each, in total 240s on vestibular and 240s on the palatal side per tooth. The treated surface was 1cm2. The power of the laser was 90mW, wavelength 660n, beam area 1 cm2, irradiance per target 0.09 W/cm2, during 240 seconds of treatment interval per point- 21.6J/cm2 of energy was delivered.
  The same laser treatment was performed the next day, as the pain was noted to be highest within 24 hours after the placement of separators.
  Other Names: LLLT

SUMMARY:
It has been reported that 90% of the patients experience pain during orthodontic treat-ment. The purpose of this study was to compare the effect of a double dose of photobio-modulation (PBM) therapy on pain perception in patients having fixed appliance treat-ment.

Twenty-two patients were recruited to participate in this single-blinded, place-bo-controlled study. Four elastomeric separators were placed, mesially and distally to the upper first molar on each side. The right side of the upper jaw was treated with low-power diode laser, and the left side was a placebo, same treatment with laser switched off. Two doses of PBM therapy (660nm, 90mW) were delivered 24 hours apart. The par-ticipants filled out the questionnaire immediately after the placement of separators and before 1st laser treatment (TO), 12 hours (T1), 24 hours (T2), 2 days (T3) and 3 days after the 1st treatment (T4). At each evaluation period, the degree of pain was scored twice, one for each side.

DETAILED DESCRIPTION:
Placing elastomeric separators is a part of the orthodontic treatment to create space for the orthodontic bands. This initial tooth displacement induces pain and instant release bio-chemical mediators such as prostaglandin-E2, substance P and interleukin 1-beta.

It has been reported that 90% of the patients experience pain in at least one part of the orthodontic treatment. Pain starts two hours after application of orthodontic fixed appliance, raises over the next 24-36 hours, starts to decrease on day 3, and disappears within 6-7 days.There are two principal groups of methods for controlling orthodontic pain: pharmacolog-ical and non-pharmacological.

Laser photobiomodulation (PBM), also called low-level laser therapy (LLLT), is the ap-plication of the light to pathology to encourage tissue regeneration, decrease inflammation and relieving pain. The wavelength used for this purpose is in the red and infrared spectrum (600-1000nm). There is no complete understanding of the mechanisms behind PBM, however enormous upturn has been done in this part. PBM has an impact on molecular, cellular and tissue level.

Past studies in this field have demonstrated the opposite outcomes of PBM therapy on relieving the pain after the insertion of orthodontic separators. Part of the researches showed a positive effect in pain reduction and some presented no effect. The studies with positive outcomes have no consistent specification such as wavelength, dose, radiant exposure, irradiance, tip diameter, average power output, peak power (for gated mode), time, or position of the points of application.

Thus, the purpose of this study was to evaluate the efficiency of low-level diode laser in decreasing the level of pain at the beginning of an orthodontic treatment caused by elas-tomeric separators. The null hypothesis for this study was that no difference existed among laser-treated and placebo side in reducing pain caused by elastomeric separators.

Materials and methods Study design This is a single-blinded, placebo-controlled, split-mouth study. The design of this study was split-mouth to eliminate all components related to differences among subjects. The study was carried out at Department of Orthodontics, University Dental Clinic, Clinical Hospital Center Rijeka. Ethical approval was obtained from the Ethical Committee of the Clinical Hospital Center of Rijeka, Croatia (003-05/2/-1-/22, 2170-29-02/1-20-2).

Sample size The sample size was decided by the Power analysis (G*power 3.1.) based on the results from the previous study [29] and predicting study power of 0.95 and a significance level of 0.05. The program calculated the sample size of at least 22 participants.

Participants and inclusion criteria The sample included 22 participants (12 females and 10 males) Procedure Four elastomeric separators (American Orthodontics, Sheboygan, WI, USA were placed, mesially and distally to the upper first molar on each side, with a specially designed plier (Hu-Friedy, Chicago, IL, USA).

Both the laser and the placebo sides were applied by the diode laser (Laser HF, Hager-Werken GmbH & Co., Duisburg, Germany), which was set at PDT mode (660nm) acu-puncture therapy. The power of the laser was set at 90 mW in intervals of 80 seconds as recommended by the manufacturer.

It was determined in advance that the right side of the upper jaw was treated with laser, and the left side was placebo.

The laser was applied perpendicular in contact with the mucosa on 1 point of the buccal and 1 point on the palatal side of the first molar approximately on the middle part of the root, with the 10mm distance from the laser to the mucosa. Each point was treated in 3 intervals, 80s each, in total 240s on vestibular and 240s on the palatal side per tooth. The treated surface was 1cm2. The power of the laser was 90mW, wavelength 660n, beam area 1 cm2, irradiance per target 0.09 W/cm2, during 240 seconds of treatment interval per point- 21.6J/cm2 of energy was delivered, with total energy applied 43.2 J per tooth. Pla-cebo side was treated the same way with the difference that the laser was switched off, but with the maintained sound signal, implying laser was working, so that participants were blinded to the allocation of the group, only the operator knew whether the side is laser treated or placebo. During the period of the laser irradiation, both the patient and orthodontist used goggles designed to block the laser's wavelength.

The same laser treatment was performed the next day, as the pain was noted to be highest within 24 hours after the placement of separators.

ELIGIBILITY:
Inclusion Criteria:

-patients aged between 12-19 years referred for orthodontic treatment, no previous orthodontic treatment, good general health , permanent dentition including second molars erupted, intact first maxillary permanent molars, good interproximal contacts on all maxillary first permanent molars, healty periodontal tissues ( gingival index=0, plaque index<1, probing depths<3mm, no peridontal attachment loss and no radiographic evidence of periodontal bone loss)

Exclusion Criteria:

* gingivitis/ periodontitis
* interproximal fillings
* missing teeth
* crowding or spacing in premolar or molar area
* severe systemic disease
* antibiotics or analgesics prescribed 15 days prior/during study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Assesment of pain | 3 days
  The pain was assessed with a visual analogue scale (VAS), which is a 100-mm-long hori-zontal line where one end corresponds to "no pain" and the other end indicates "worst pain possible." The participants filled out the questionnaire immediately after the placement of separators (TO) and before 1st laser treatment, 12 hours (T1), 24hours (T2) and just after 2nd laser treatment, 2 days (T3) and 3 days after the 1st treatment (T4) (Table 1). At each evalua-tion period, the degree of pain was scored twice, one for each side. Each patient was re-quired to indicate whether he/she had taken any analgesics during the recorded period.

CONTACTS AND LOCATIONS:
Overall Officials: Senka Mestrovic, DDS, PhD, Study Director — University of Zagreb
Locations (1):
- University Hospital Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No